CLINICAL TRIAL: NCT01769729
Title: Program for Emotional and Physical Pain - Pilot Randomized Clinical Trial
Acronym: PEPP - RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MH085762; R34MH085762 (NIH)
Record Dates: First submitted 2013-01-15; First posted 2013-01-17 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Depression; Chronic Low Back Pain
Keywords: integrated primary care; depression; chronic low back pain
MeSH Terms: conditions — Depression | interventions — CDRI 85-287

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PEPP + care management (Experimental): This 4-month collaborative psychotherapy, entitled Program for Emotional and Physical Pain (PEPP), will include 1 joint meetings with the behavioral health specialist (BHS), primary care provider (PCP), and patient, 10 psychotherapy sessions, and continued collaboration between the BHS and the PCP to assure a shared treatment plan.
  Care management will include monthly calls with a depression care manager.
  Interventions: Behavioral: PEPP; Behavioral: Care management
- Care management alone (Active Comparator): Care management will include monthly calls with a depression care manager.
  Interventions: Behavioral: Care management

INTERVENTIONS:
Behavioral: PEPP
  Arms: PEPP + care management
Behavioral: Care management

SUMMARY:
The overall aim of this program of research is to develop a collaborative psychotherapy for major depressive disorder (MDD) specifically for primary care patients with MDD and comorbid chronic low back pain (CLBP).

The purpose of the proposed project is to establish the feasibility and acceptability of a research design for an eventual large-scale randomized clinical trial which would test the efficacy of PEPP in comparison to a control condition (depression care management).

To achieve the investigators specific aims, the investigators will conduct a pilot randomized clinical trial (n = 30), with two treatment arms; PEPP (which includes procedures used in care management) or care management.

DETAILED DESCRIPTION:
The overall aim of this program of research is to develop a collaborative psychotherapy for major depressive disorder (MDD) specifically for primary care patients with MDD and comorbid chronic low back pain (CLBP). The newly developed intervention will integrate and build on behavior therapy for MDD and behavior therapy for chronic pain towards a key target of reducing behavioral avoidance. This 4-month collaborative psychotherapy, entitled Program for Emotional and Physical Pain (PEPP), will include 1 joint meeting with the behavioral health specialist (BHS), primary care provider (PCP), and patient, 10 psychotherapy sessions, and continued collaboration between the BHS and the PCP to assure a shared treatment plan.

The purpose of the proposed project is to establish the feasibility and acceptability of a research design for an eventual large-scale randomized clinical trial which would test the efficacy of PEPP in comparison to a control condition (depression care management)..

To achieve the investigators specific aims, the investigators will conduct a pilot randomized clinical trial (n = 30), with two treatment arms; PEPP (which includes procedures used in care management) or care management. The specific aims are:

1. To develop and refine PEPP so that it meets standards of feasibility and acceptability for primary care physicians (PCPs), behavioral health specialists (BHSs), and participants;

   1. To develop, field-test, and finalize a PEPP manual;
   2. To develop a reliable measure of BHS adherence to the manual;
   3. To develop, field-test, and finalize BHS training and supervision procedures;
2. To field-test and finalize procedures for depression care management;
3. To establish that the investigators can adequately provide depression care management and that it is acceptable in this population;
4. To develop and refine recruitment methods for an RCT and document an adequate rate of recruitment;
5. To refine research procedures, e.g., consent process, randomization process, and assessment procedures, and establish their feasibility and acceptability to participants.

Ultimately, the investigators expect that this treatment development work will prepare us to apply for an R01 to conduct a large-scale, adequately powered RCT with the same research design as the pilot RCT proposed in this application. Depression will be the primary outcome variable assessed in the large-scale RCT; pain will be a secondary outcome variable. In the end, the investigators believe this line of work will lead to the incorporation into primary care of theoretically-driven and effective mental health treatment for patients with MDD and comorbid CLBP. To the best of the investigators knowledge, this would be the first empirically-tested psychotherapy protocol that specifically integrates treatment of major depression with CLBP.

ELIGIBILITY:
Inclusion Criteria:

1. Meets DSM-IV criteria for current major depressive disorder.
2. Participants must have a Quick Inventory of Depressive Symptoms (QIDS) score >11.
3. Chronic low back pain. Pain must be > 6 months duration, in the low back (lumbar region), present > ½ the days of the month, and, on average, be of at least a moderate level of severity in the last month (> 4 on an 11-point numerical rating of pain intensity ranging from 0 [no pain] to10 [worst pain imaginable]. Pain-related disability / functional impact of pain must be of at least moderate severity at the time of intake, determined by a score of at > 7 on the Roland Morris Disability Questionnaire (RMDQ; (Roland & Morris, 1983))
4. Continued pain despite having attempted initial steps of PCP guideline-based care (Chou et al., 2007). Participants must have been under the care of a physician for low back pain for > 6 months and have already had > 2 trials of recommended medications (i.e., acetaminophen, NSAIDs, skeletal muscle relaxants, opioids, and/or benzodiazepines).This will be judged through chart review and interviews with patients & PCPs.
5. Antidepressant dose stable for previous 2 months. If the participant is taking an antidepressant, he/ she must have been on the same dose for the previous 2 months.
6. Aged 18 or older.
7. Have a PCP at one of our enrollment sites.

Exclusion Criteria:

1. Lifetime diagnosis of bipolar disorder, schizophrenia, or other chronic psychotic condition.
2. Current hazardous illicit drug or alcohol use assessed with the AUDIT and DUDIT.
3. Opiate misuse will be assessed with the COMM and via primary care chart review.
4. Suicidal ideation or behavior requiring immediate attention.
5. In psychotherapy or in a multidisciplinary pain management program at baseline.
6. Anticipate having surgery in the next 6 months.
7. Pain thought to be due to visceral disease, cancer, infection, or inflammatory arthritis or pain associated with severe or progressive neurological deficits.
8. Current pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Quick Inventory of Depression Symptoms | 4 months
  assessment of depression

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Uebelacker, PhD, Principal Investigator — Butler Hospital, Brown University; Risa Weisberg, PhD, Principal Investigator — Brown University
Locations (1):
- Family Care Center of Memorial Hospital, Pawtucket, Rhode Island, United States